CLINICAL TRIAL: NCT06072742
Title: Effect of Lifestyle on Caries and Apical Periodontitis: Results From a University-based Cross-sectional Study
Brief Title: Effect of Lifestyle on Caries and Apical Periodontitis
Status: Completed | Type: Observational
Sponsor: University of Siena (Other)
Responsible Party: Principal Investigator, Simone Grandini, Professor, University of Siena
Other Study IDs: LS002
Record Dates: First submitted 2023-10-02; First posted 2023-10-10 (Actual); Last update posted 2023-12-01 (Actual); Status verified 2023-11

CONDITIONS: Apical Periodontitis; Caries; Lifestyle; Inflammation; Endodontics
Keywords: Apical periodontitis; caries; inflammation; Endodontics; lifestyle
MeSH Terms: conditions — Periapical Periodontitis; Inflammation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study aimed to link lifestyle factors (Mediterranean diet adherence, stress, sleep quality, physical activity) to caries and apical periodontitis in 149 university-based individuals. Data included clinical and radiographic assessments and lifestyle questionnaires. Statistical tests and logistic regression were employed to analyze the relationships between these factors and oral health conditions.

DETAILED DESCRIPTION:
The aim of this study was to evaluate the association between lifestyle (adherence to the Mediterranean diet, stress, sleep quality, and level of physical activity) with the presence of caries and apical periodontitis (AP) in a University-based cohort of individuals.

A total of 149 patients were included in this cross-sectional study. In addition to clinical (cold test, percussion test, evaluation of tooth mobility) and radiographic (bitewing Rx, periapical Rx, and OPT) parameters, validated questionnaires were used to investigate patient's lifestyle. Data on the number of decayed, missing, and filled teeth (DMFT score) and the severity of apical periodontitis (PAI score) were extrapolated from the available clinical and instrumental investigations. Shapiro-Wilk test was used to evaluate the normal distribution of data; Wilcoxon rank-sum test (Mann-Whitney) was used to compare continuous variables. Fisher's test was used to compare dichotomized variables. A logistic regression model was performed for the multivariate analysis.

ELIGIBILITY:
Inclusion Criteria:

* age between 18 and 70
* Good general health status;
* Ability and willingness to give written consent;
* Presence of at least 6 teeth.

Exclusion Criteria:

* Age <18 years;
* Pregnancy or lactation;
* administration of antibiotics within the last 6 months;
* Inability and unwillingness to give written consent

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All consecutive patients attending the Unit of Endodontics at the University of Siena were screened between September 2020 and August 2021. Patients were eligible based on the inclusion criteria. Individuals were included in the study after they read and signed the written informed consent, in accordance with the Declaration of Helsinki.
Sampling Method: Non-Probability Sample
Enrollment: 149 (Actual)
Dates: Start 2020-09-20 (Actual); Primary Completion 2021-08-20 (Actual); Study Completion 2021-08-20 (Actual)

PRIMARY OUTCOMES:
Presence of Apical Periodontitis | The time frame for this observational study is defined by the initial assessment conducted at baseline. No follow-up measurements are scheduled, and the study aims to explore associations and characteristics at a single time point
  The periapical status was investigated by palpation, percussion, thermal cold testing, and panoramic radiographs. Afterward, teeth that exhibited deep carious lesions, deep restorations, no response to pulp testing, or painful response to biting and/or percussion or palpation were suspected of AP. Those teeth underwent further periapical radiograph using the long cone paralleling technique with a film holder. AP cases were diagnosed based on the identification of at least one tooth with periapical radiolucency outpacing twice the width of the periodontal ligament space and having PAI > 2.
Periapical index (PAI) | The time frame for this observational study is defined by the initial assessment conducted at baseline. No follow-up measurements are scheduled, and the study aims to explore associations and characteristics at a single time point
  Periapical health was assessed radiographically using the PAI score that was determined through visual inspection of the periapical area, assigning a numerical value based on the extent and severity of inflammation. Scores ranged from 0 to 5
Decayed, missing, filled teeth (DMFT) index | The time frame for this observational study is defined by the initial assessment conducted at baseline. No follow-up measurements are scheduled, and the study aims to explore associations and characteristics at a single time point
  The DMFT index is calculated by summing the scores for decayed (D), missing (M), and filled (F) teeth for an individual or a group of individuals

CONTACTS AND LOCATIONS:
Overall Officials: Simone Grandini, DDS, Study Director — University of Siena
Locations (1):
- Azienda Ospedaliera Universitaria Senese, Siena, Italy

IPD SHARING:
Plan to Share IPD: Undecided
no plan to share IPD